CLINICAL TRIAL: NCT03440411
Title: A MULTICENTER, OPEN LABEL, RANDOMIZED PHASE III STUDY OF POMALIDOMIDE-DEXAMETHASONE vs POMALIDOMIDE-CYCLOPHOSPHAMIDE-DEXAMETHASONE IN MULTIPLE MYELOMA (MM) PATIENTS WHO EXPERIENCE BIOCHEMICAL OR CLINICAL RELAPSE DURING LENALIDOMIDE MAINTENANCE TREATMENT
Brief Title: Pom-dex Versus Pom-Cyclo-dex in MM Patients With Biochemical or Clinical Relapse, During Lena Maintenance Treatment
Acronym: PO-3887
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: PO-CL-MM-PI-003887
Record Dates: First submitted 2018-02-07; First posted 2018-02-22 (Actual); Results first posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Multiple Myeloma
Keywords: biochemical relapse
MeSH Terms: conditions — Multiple Myeloma | interventions — pomalidomide; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: This is a 2x2 factorial randomized study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ARM pom-dex Early (A-I) (Active Comparator): Patients will receive treatment at biochemical relapse with pom-dex Pomalidomide: 4 mg/day on days 1-21 Dexamethasone: 40 mg on days 1, 8, 15, 22 For 28-day cycles until progression or intolerance
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- ARM pom-cyclo-dex Early(B-I) (Experimental): Patients will receive treatment at biochemical relapse with pom-cyclo-dex Pomalidomide: 4 mg/day on days 1-21 Cyclophosphamide: 50 mg every other day Dexamethasone: 40 mg on days 1, 8, 15, 22 For 28-day cycles until progression or intolerance
  Interventions: Drug: Pomalidomide; Drug: Cyclophosphamide; Drug: Dexamethasone
- ARM pom-dex Late (A-II) (Experimental): Patients will be randomized at biochemical relapse and they will start treatment with pom-dex at the onset of CRAB symptoms/significant paraprotein increase.
  Pomalidomide: 4 mg/day on days 1-21 Dexamethasone: 40 mg on days 1, 8, 15, 22 For 28-day cycles until progression or intolerance
  Interventions: Drug: Pomalidomide; Drug: Dexamethasone
- ARM pom-cyclo-dex Late (B-II) (Active Comparator): Patients will be randomized at biochemical relapse and they will start treatment with pom-cyclo-dex at the onset of CRAB symptoms/significant paraprotein increase.
  Pomalidomide: 4 mg/day on days 1-21 Cyclophosphamide: 50 mg every other day Dexamethasone: 40 mg on days 1, 8, 15, 22 For 28-day cycles until progression or intolerance
  Interventions: Drug: Pomalidomide; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Pomalidomide — 4 mg/daily as oral administration (PO) on days 1-21.
  Other Names: Imnovid(R)
Drug: Cyclophosphamide — 50 mg every other day as oral administration (PO) on days 1-28
  Other Names: Endoxan(R)
  Arms: ARM pom-cyclo-dex Early(B-I); ARM pom-cyclo-dex Late (B-II)
Drug: Dexamethasone — 40 mg as oral administration (PO) on days 1, 8, 15, 22.
  Other Names: Soldesam(R)

SUMMARY:
The combination lenalidomide plus low-dose dexamethasone (Rd) is an active treatment for Multiple Myeloma (MM) patients, both at diagnosis and at relapse.

Pomalidomide, is an immunomodulatory molecule (IMID), derivative of thalidomide, developed to improve the efficacy and reduce the toxicity of the parent molecule. Pomalidomide and dexamethasone (pom-dex) proved to be an effective and safe treatment in MM patients refractory to lenalidomide and refractory/intolerant to bortezomib.

The addition of chemotherapy to novel drugs has been evaluated both at diagnosis and at relapse. The combination of pomalidomide-cyclophosphamide-prednisone proved to be safe and effective in relapsed/refractory MM patients. The combination pomalidomide-cyclophosphamide-dexamethasone (pom-cyclo-dex) was tested in a phase II study in patients with relapsed and refractory MM, demonstrating a good tolerability using pomalidomide at the dose of 4 mg. Pom-cyclo-dex resulted in a superior response rate and Progression-Free Survival (PFS) compared to pom-dex. The increased hematologic toxicities, as a result of the addition of oral cyclophosphamide, were manageable. With an overall response rate of 65% the combination demonstrated a promising efficacy.The first aim of our trial, is to compare the combination of pom-cyclo-dex vs pom-dex.

Relapsed myeloma is defined as previously treated myeloma that progresses and requires the initiation of salvage therapy.

According to International Myeloma Working Group (IMWG) recommendation, biochemical relapse is defined as an increase of ≥ 25% of tumor burden from lowest value, without any CRAB feature (CRAB is defined as the onset of clinical symptoms: hypercalcemia, renal failure, anemia and bone lesions) and detected in 2 consecutive determinations.

Clinical relapse requires one or more direct indicators of progressive disease and end organ dysfunction (CRAB features).

Treatment at relapse should start in case of clinical relapse or a significant paraprotein increase (doubling of M-component in 2 months).

In case of biochemical relapse the standard is observation only, as in case of asymptomatic MM at diagnosis.

However, a recently published trial, showed improved PFS and OS for newly diagnosed asymptomatic patients treated with lenalidomide and dexamethasone in comparison with observation only. Our hypothesis is that similarly, in the relapse setting, patients may benefit from an early intervention, meaning a treatment at biochemical relapse and not only in case of clinical relapse or rapid increase of M-component.

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a neoplastic disease of older adults, with a higher incidence in elderly patients: 26% are aged 65-74 years, and 37% are older than 75 years. The annual prevalence of MM is approximately 31 cases per 100,000 people in patients aged 65-74 years, and it increases to 46 cases per 100,000 people in patients aged ≥75 years. The prevalence of myeloma is likely to increase due to the extended survival and the growing life expectancy of the general population.

Recently, the introduction of novel agents such as thalidomide, lenalidomide, pomalidomide and bortezomib, has changed the treatment paradigm of MM and extended survival.

The prognosis of patients who are refractory to novel agents is especially poor. A retrospective study has recently demonstrated that patients with relapsed MM, who were refractory to bortezomib and were relapsed following, refractory to or ineligible to receive treatment with an IMiD, had a median overall survival (OS) and event free survival (EFS) of 9 and 5 months, respectively.

STUDY DESIGN When patients experience biochemical relapse during lenalidomide maintenance, they will stop lenalidomide, as established in the related experimental protocol. Afterwards, patients can be considered for the enrollment in the present study if all inclusion and exclusion criteria are met.

This is a multicenter, randomized, open label phase III study designed to assess the safety and the efficacy of two different pomalidomide combinations as salvage treatment in multiple myeloma (MM) patients.

Patients will be evaluated at scheduled visits in up to 3 study periods: pre-treatment, treatment and long-term follow-up (LTFU).

The pre-treatment period includes screening visits, performed at study entry. After providing written informed consent to participate in the study, patients will be evaluated for study eligibility. The screening period includes the availability of inclusion criteria described above.

The treatment period includes administration of pomalidomide and dexamethasone in arm A and pomalidomide combined with cyclophosphamide and dexamethasone in arm B. The response will be assessed after each cycle. Patients will be randomized to receive treatment at biochemical relapse (ARM I) or at clinical relapse (ARM II).

The LTFU periods will start after development of confirmed progression disease (PD), all patients are to be followed for survival during the LTFU period every 3 months via telephone or office visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years and <80 years.
* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Male patient agrees to use an acceptable method for contraception (i.e. condom or abstinence) for the duration of the study.

Female of childbearing potential agrees to use two acceptable methods for contraception [implant, levonorgestrel-releasing intrauterine system (IUS), medroxyprogesterone acetate depot, tubal sterilization, sexual intercourse with a vasectomised male partner only (vasectomy must be confirmed by two negative semen analyses), ovulation inhibitory progesterone-only pills (i.e. desogestrel)] or absolute and continuous sexual abstinence.

* Patient has measurable disease, defined as follows: any quantifiable serum monoclonal protein value (generally, but not necessarily, ≥ 0.5 g/dL of M-protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours; only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved Free Light Chain (FLC) levels must be > 10 mg/dL. Less than 10% of oligo- or non-secretory MM patients with free light chains will be admitted to this study in order to maximize interpretation of benefit results.
* Patient receiving lenalidomide maintenance therapy as part of first line treatment (concomitant use of prednisone is accepted) and has experienced a biochemical relapse, with evidence of progressive disease defined as an increase of 25% from lowest response value in any one or more of the following: serum M-component (absolute increase must be ≥0.5 g/100 ml) and/or urine M-component (absolute increase must be ≥200 mg per 24 hours) only in patients without measurable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels must be >10 mg/dL (35).
* Patient who received as first line treatment a bortezomib-based therapy, including lenalidomide maintenance during the same line of therapy, can be included in the trial.
* Patient has a life-expectancy > 3 months
* Patient has not a currently active malignancy, other than non melanoma skin cancer and carcinoma in situ of the cervix, and has not invasive malignancies within the past 5 years.
* No history of allergic reactions attributed to study agents
* Patient has the following laboratory values within 28 days before baseline day 1 of the cycle 1:

  1. absolute neutrophil count (ANC) > 1 x 10^9/L
  2. platelet count > 75 x 10^9/L
  3. haemoglobin > 8 g/dl.
  4. aspartate transaminase (AST): < 2 x the upper limit of normal (ULN).
  5. alanine transaminase (ALT): < 2 x the ULN.

Exclusion Criteria:

* Pregnant or lactating females.
* Patient with Creatinine Clearance (CrCl) < 45 mL/minute
* Patient with peripheral neuropathy ≥ Grade 2
* Subject with any one of the following:
* Congestive heart failure (NY Heart Association Class III or IV)
* Myocardial infarction within 12 months prior to starting study treatment
* Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris
* Any significant medical disease or conditions (e.g. pulmonary disease, infection) that, in the investigator's opinion, may interfere with protocol adherence or subject's ability to give informed consent or could place the subject at unacceptable risk.
* Clinical active infectious hepatitis type A, B, C or HIV Acute active infection requiring antibiotics or infiltrative pulmonary disease
* Contraindication to any of the required drugs or supportive treatments.
* Known allergy to any of the study medications, their analogues, or excipients in the various formulations

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-02-18 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione EMN Italy Onlus, Torino, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At enrollment patients was randomized to receive Late (II) vs Early (I) treatment and Pom-Cyclo-dex (B) vs Pom-dex (A) at the same time. If patient was randomized to receive I treatment, the result of the comparison between BvsA was immediately available. Otherwise, in case of II treatment the random disclosure of the comparison between B vs A arm was at the confirmation of CRAB. Patients was randomized using blocks of sizes 12 by the electronic Case Report Form.
Pre-assignment Details: For previous reason 1pt randomized to Late (II) treatment who not achieved a CRAB has not the disclosure of the randomization between A vs B arm.
Groups:
- ARM Pom-dex Early (A-I): Patients will receive treatment at biochemical relapse with pom-dex Pomalidomide: 4 mg/daily as oral administration (PO) on days 1-21. Dexamethasone: 40 mg as oral administration (PO) on days 1, 8, 15, 22. For 28-day cycles until progression or intolerance
- ARM Pom-dex Late (A-II): Patients will be randomized at biochemical relapse and they will start treatment with pom-dex at the onset of CRAB symptoms/significant paraprotein increase.
  Pomalidomide: 4 mg/daily as oral administration (PO) on days 1-21. Dexamethasone: 40 mg as oral administration (PO) on days 1, 8, 15, 22. For 28-day cycles until progression or intolerance
- ARM Pom-cyclo-dex Early (B-I): Patients will receive treatment at biochemical relapse with pom-cyclo-dex Pomalidomide: 4 mg/daily as oral administration (PO) on days 1-21. Cyclophosphamide: 50 mg every other day as oral administration (PO) on days 1-28 Dexamethasone: 40 mg as oral administration (PO) on days 1, 8, 15, 22. For 28-day cycles until progression or intolerance
- ARM Pom-cyclo-dex Late (B-II): Patients will be randomized at biochemical relapse and they will start treatment with pom-cyclo-dex at the onset of CRAB symptoms/significant paraprotein increase.
  Pomalidomide: 4 mg/daily as oral administration (PO) on days 1-21. Cyclophosphamide: 50 mg every other day as oral administration (PO) on days 1-28 Dexamethasone: 40 mg as oral administration (PO) on days 1, 8, 15, 22. For 28-day cycles until progression or intolerance
Period: Overall Study
Arm/Group | ARM Pom-dex Early (A-I) | ARM Pom-dex Late (A-II) | ARM Pom-cyclo-dex Early (B-I) | ARM Pom-cyclo-dex Late (B-II)
Started | 3 | 1 | 2 | 2
Completed (Treatment is continous until progression disease (PD), so treatment has not a specific duration and so "completed" is Not Applicable.) | 0 | 0 | 0 | 0
Not Completed | 3 | 1 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — PD | 2 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Closed study by sponsor | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: This analysis included only patients in whom CPd vs Pd randomization was disclosed; 1pt randomized to Late (II) treatment who not achieved a CRAB has not the disclosure of the randomization between A vs B arm..
Groups:
- Total: Total of all reporting groups
Arm/Group | ARM Pom-dex Early (A-I) | ARM Pom-dex Late (A-II) | ARM Pom-cyclo-dex Early (B-I) | ARM Pom-cyclo-dex Late (B-II) | Total
Number analyzed (Participants) | 3 | 1 | 2 | 2 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 1 | 2 | 5
  >=65 years | 1 | 1 | 1 | 0 | 3
Age, Continuous [Median (Full Range); unit: years] | 54 [43 to 79] | 68 [68 to 68] | 59.5 [52 to 67] | 60 [60 to 60] | 60 [43 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 0 | 2
  Male | 2 | 1 | 1 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 3 | 1 | 2 | 2 | 8
Region of Enrollment [Number; unit: participants]
  Italy | 3 | 1 | 2 | 2 | 8
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — ECOG 0-5; the best is 0, 5 is death
  participants
    0 | 2 | 0 | 1 | 2 | 5
    1 | 1 | 1 | 1 | 0 | 3
isotype [Count of Participants; unit: Participants]
  IgG | 3 | 0 | 2 | 2 | 7
  Bj | 0 | 1 | 0 | 0 | 1
International Staging System (ISS) Stage [Count of Participants; unit: Participants] — International Staging System (ISS) for Multiple Myeloma Stage VALUES (β2M = Serum β2 microglobulin; ALB = serum albumin I β2M < 3.5 mg/L; ALB ≥ 3.5 g/dL II β2M < 3.5 mg/L; ALB ≥ 3.5 g/dL; or β2M 3.5 - 5.5 mg/L III β2M > 5.5 mg/L I low risk, II medium risk, III high risk
  Participants
    I | 2 | 0 | 2 | 2 | 6
    II | 1 | 1 | 0 | 0 | 2
Previous Therapies (induction/Autologous Stem Cell Transplantation/consolidation) [Count of Participants; unit: Participants]
  ASCT | 2 | 1 | 2 | 2 | 7
  Len | 3 | 0 | 2 | 2 | 7
  Bort | 2 | 0 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: defined as the time from the date of random disclosure to the date of death from any cause for the comparisons B vs A
Time Frame: 57 months
Population: This analysis included only patients in whom CPd vs Pd randomization was disclosed.
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Pd
- Arm B: CPd
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 4 | 4
Participants
  Death | 2 | 0
  Censored | 2 | 4

2. Primary Outcome: Overall Survival
Description: defined as the time from the date of random disclosure to the date of death from any cause for the comparisons II vs I
Time Frame: 57 months
Population: This analysis included only patients in whom CPd vs Pd randomization was disclosed.
Measure: Count of Participants; unit: Participants
Groups:
- Arm I: Early Treatment
- Arm II: Late treatment
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 5 | 3
Participants
  Death | 1 | 1
  Censored | 4 | 2

3. Secondary Outcome: Clinical Progression
Description: defined as the time from random assignment to the early or late strategy to the date of onset of CRAB symptoms or death.
  Clinical relapse requires one or more direct indicators of progressive disease and end organ dysfunction (CRAB features). Evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder:
  * hypercalcaemia
  * renal insufficiency
  * anaemia
  * bone lesions
  Any one or more of the following biomarkers of malignancy:
  * clonal bone marrow plasma cell percentage ≥60%
  * involved:uninvolved serum free light chain ratio ≥100
  * >1 focal lesions on MRI studies (each focal lesion must be 5 mm or more in size)
  Progresson was defined accoring to IMWG criteria as reported before
Time Frame: 57 months
Population: All population
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 5 | 4
Participants
  Not evaluable | 5 | 3
  Without CRAB | 0 | 1

4. Secondary Outcome: Progression Free-survival (PFS)
Description: PFS for the comparison B vs A will be measured from the date of randomization disclosure to the date of first observation of PD, or death from any cause as an event. Subjects who have not progressed or who withdraw from the study will be censored at the time of the last complete disease assessment. All subjects who were lost to Follow Up (FU) will also be censored at the time of last complete disease assessment
Time Frame: 57 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 4 | 4
Participants
  Events | 3 | 1
  Censored | 1 | 3

5. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS for the comparison II vs I will be measured from the date of randomization disclosure to the date of first observation of PD, or death from any cause as an event. Subjects who have not progressed or who withdraw from the study will be censored at the time of the last complete disease assessment. All subjects who were lost to FU will also be censored at the time of last complete disease assessment
Time Frame: 57 months
Population: This analysis included only patients in whom CPd vs Pd randomization was disclosed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 5 | 3
Participants
  Events | 3 | 1
  Censored | 2 | 2

6. Secondary Outcome: Progression Free-survival 2(PFS2)
Description: PFS for the comparison B vs A will be measured from the date of randomization disclosure to the date of first observation of PD in second line therapy, or death from any cause as an event. Subjects who have not progressed or who withdraw from the study will be censored at the time of the last complete disease assessment. All subjects who were lost to FU will also be censored at the time of last complete disease assessment
Time Frame: 57 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 4 | 4
Participants
  Events | 2 | 1
  Censored | 2 | 3

7. Secondary Outcome: Progression Free Survival 2(PFS2)
Description: PFS for the comparison II vs I will be measured from the date of randomization disclosure to the date of first observation of PD in second line therapy, or death from any cause as an event. Subjects who have not progressed or who withdraw from the study will be censored at the time of the last complete disease assessment. All subjects who were lost to FU will also be censored at the time of last complete disease assessment
Time Frame: 57 months
Population: This analysis included only patients in whom CPd vs Pd randomization was disclosed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 5 | 3
Participants
  Events | 2 | 1
  Censored | 3 | 2

8. Secondary Outcome: Objective Overall Response Rate for the Comparison B vs A
Description: in terms of partial response (PR), very good partial response (VGPR), complete response (CR).and stringent complete response (sCR) according to IMWG response crieria (https://www.myeloma.org/resource-library/international-myeloma-working-group-imwg-uniform-response-criteria-multiple).
Time Frame: 57 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 4 | 4
Participants
  sCR | 0 | 0
  CR | 0 | 0
  VGPR | 0 | 0
  PR | 0 | 3
  SD | 2 | 0
  PD | 1 | 1
  NE | 1 | 0

9. Secondary Outcome: Objective Overall Response Rate for the Comparison II vs I
Description: as for outcome 8
Time Frame: 57 months
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 5 | 3
Participants
  sCR | 0 | 0
  CR | 0 | 0
  VGPR | 0 | 0
  PR | 1 | 2
  SD | 2 | 0
  PD | 1 | 1
  NE | 1 | 0

10. Secondary Outcome: Quality of Life Questionnaire (QLQ) With EORTC-QLQ-C30
Description: outcome will be measured with EORTC-QLQ-C30 at baseline, every 2 months during the first year, and then every 6 months for the comparison B vs B and I vs II.
Time Frame: 57 months
Population: data could not be reported in the data table since analysis was not performed according to the lower sample size and QLQ missing
Groups:
- ARM A-I: Patients will receive treatment at biochemical relapse with pom-dex Pomalidomide: 4 mg/daily as oral administration (PO) on days 1-21. Dexamethasone: 40 mg as oral administration (PO) on days 1, 8, 15, 22. For 28-day cycles until progression or intolerance
- ARM A-II: Patients will be randomized at biochemical relapse and they will start treatment with pom-dex at the onset of CRAB symptoms/significant paraprotein increase.
  Pomalidomide: 4 mg/daily as oral administration (PO) on days 1-21. Dexamethasone: 40 mg as oral administration (PO) on days 1, 8, 15, 22. For 28-day cycles until progression or intolerance
- ARM B-I: Patients will receive treatment at biochemical relapse with pom-cyclo-dex Pomalidomide: 4 mg/daily as oral administration (PO) on days 1-21. Cyclophosphamide: 50 mg every other day as oral administration (PO) on days 1-28 Dexamethasone: 40 mg as oral administration (PO) on days 1, 8, 15, 22. For 28-day cycles until progression or intolerance
- ARM B-II: Patients will be randomized at biochemical relapse and they will start treatment with pom-cyclo-dex at the onset of CRAB symptoms/significant paraprotein increase.
  Pomalidomide: 4 mg/daily as oral administration (PO) on days 1-21. Cyclophosphamide: 50 mg every other day as oral administration (PO) on days 1-28 Dexamethasone: 40 mg as oral administration (PO) on days 1, 8, 15, 22. For 28-day cycles until progression or intolerance
Arm/Group | ARM A-I | ARM A-II | ARM B-I | ARM B-II
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Quality of Life With QLQ-MY(Myeloma)24
Description: outcome will be measured with QLQ-MY24 at baseline, every 2 months during the first year, and then every 6 months for the comparison B vs B and I vs II.
Time Frame: 57 months
Population: as for outcome 10
Arm/Group | ARM A-I | ARM A-II | ARM B-I | ARM B-II
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: from randomization through study completion, up to 57 months, an average of 45 months
Description: In the table "Other Adverse Events" each term reports ae term_ctcae grade
Arm/Group | ARM Pom-dex Early (A-I) | ARM Pom-dex Late (A-II) | ARM Pom-cyclo-dex Early (B-I) | ARM Pom-cyclo-dex Late (B-II)
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/1 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/1 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/3 | 1/1 | 1/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM Pom-dex Early (A-I) (N=3) | ARM Pom-dex Late (A-II) (N=1) | ARM Pom-cyclo-dex Early (B-I) (N=2) | ARM Pom-cyclo-dex Late (B-II) (N=2)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ARM Pom-dex Early (A-I) (N=3) | ARM Pom-dex Late (A-II) (N=1) | ARM Pom-cyclo-dex Early (B-I) (N=2) | ARM Pom-cyclo-dex Late (B-II) (N=2)
Agitation_1 (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Agitation_2 (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Agitation_3 (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ALT increased_2 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia_1 (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AST increased_1 (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection_2 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Chills_1 (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusion_2 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation_1 (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhea_2 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme_2 (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye burns_2 (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue_1 (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue_2 (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue_3 (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Fever_3 (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flu like symptoms_2 (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis_1 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis_2 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia_2 (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension_1 (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia_2 (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leg ulcer_2 (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection_2 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung nodule_3 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle cramps_1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle cramps_3 (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness_3 (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia_3 (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (5) | 0 (0)
Pain in limb_1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in limb_2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in limb_3 (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy_2 (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope_2 (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular_2 (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia_3 (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence_2 (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superficial thrombophlebitis_2 (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia_1 (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic ulcer_3 (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection_2 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vomiting_2 (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Main limitations is that the sample size of participants needed to achieve target power and statistically reliable results was not reach. And no statistical testing was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT03440411/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-13): https://cdn.clinicaltrials.gov/large-docs/11/NCT03440411/SAP_001.pdf